CLINICAL TRIAL: NCT05561075
Title: Evaluation of the Oral Bioavailability of Pterostilbene Cocrystal Compared to Its Free Form in Healthy Volunteers. Crossover, Randomized, Double-Blind Study (BIOPTERO)
Brief Title: Oral Bioavailability of Pterostilbene Cocrystal Compared to Its Free Form (BIOPTERO)
Acronym: BIOPTERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Circe, S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: BIOPTERO
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Biological Availability
Keywords: Polyphenols; Antioxidant activity; Co-crystallization; Pterostilbene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pterostilbene cocrystal (Experimental)
  Interventions: Dietary Supplement: Pterostilbene cocrystal
- Pterostilbene free form (Active Comparator)
  Interventions: Dietary Supplement: Pterostilbene free form

INTERVENTIONS:
Dietary Supplement: Pterostilbene cocrystal — One capsule with Pterostilbene cocrystal
  Arms: Pterostilbene cocrystal
Dietary Supplement: Pterostilbene free form — One capsule with Pterostilbene free form
  Arms: Pterostilbene free form

SUMMARY:
Oxidative stress and reactive oxygen species (ROS) can seriously affect cells, tissues and organs. The human body is capable of counteracting ROS production by stimulating antioxidant defense systems and consequently adapting to the oxidative challenge.

Several transcription factors are involved in the induction of antioxidant genes. Activators of nuclear factor derived from erythroid 2 (NRF2), a protein that controls the expression of certain genes, are considered agents capable of inducing antioxidant capacity and to alleviate ROS. There are some food bioactive compounds, including polyphenols, capable of activating NRF2.

Pterostilbene (PT) is a stilbenoid found in many natural sources, and is emerging as an antioxidant due to its potential preventive and therapeutic properties in a long list of diseases. Despite its apparent properties, the water solubility and bioavailability of PT are low.

The co-crystallization of nutraceuticals is a recent strategy based on crystal engineering to overcome their low solubility and, therefore, their low oral bioavailability. It has been identified and characterized a cocrystal of pterostilbene that can increase oral bioavailability in animals by up to 10 times compared to the commercial free base PT.

The main objective of the study is to evaluate the oral bioavailability of the crystallized form of pterostilbene (ccPT) compared to its commercial free base form (pterostilbene (PT).

The secondary objectives of the study are to determine the pharmacokinetic parameters:

* Relative oral bioavailability (Frel)
* Maximum concentration (Cmax).
* Maximum time (Tmax).
* Half life time (T1/2).

During the study there will be 3 visits: a preselection visit (V0), a visit for the first postprandial study (V1) and after one week washing period, a visit for the second postprandial study (V2).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 65 years of age.
* Sign the informed consent form.
* Know how to read, write and speak Spanish

Exclusion Criteria:

* Take supplements or multivitamin supplements or phytotherapeutic products (especially infusions) that interfere with the treatment under study up to 30 days before the start of the study.
* Be lacto-vegetarian, lacto-ovo-vegetarian, or vegan.
* Present intolerances and/or food allergies related to pterostilbene.
* Be a smoker.
* Having received antibiotic treatment up to 30 days before the start of the study.
* Present values of body mass index ≤ 18kg/m^2 or ≥ 35 kg/m^2.
* Present some chronic disease with clinical manifestations: coronary heart disease, cardiovascular disease, diabetes, celiac disease, Crohn's disease, chronic kidney disease, cancer, autoimmune diseases (such as fibromyalgia), respiratory and/or gastrointestinal diseases that may compromise the absorption of the compound.
* Clinical history of anemia.
* Being pregnant or intending to became pregnant.
* Be in breastfeeding period.
* Being unable to follow the study guidelines.
* Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days before inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Pterostilbene calculated by area under the curve (AUC 0-24) of plasma pterostilbene levels. | At week 1 and week 2
  Fasting pterostilbene levels in plasma will be determined before consume the capsule with pterostilbene until 24 hours postprandially at 8 points after consuming the capsule (0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours and 24 hours).

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | At week 1 and week 2
  Maximum plasma concentration of pterostilbene
Time for maximum plasma concentration (Tmax) | At week 1 and week 2
  Time period for the maximum plasma concentration of pterostilbene.
Half-life (T1/2). | At week 1 and week 2
  Time taken for half the initial dose of pterostilbene administered to be eliminated from the body
Area Under the Curve (AUC 0-inf) of plasma pterostilbene levels. | At week 1 and week 2
  Fasting pterostilbene levels in plasma will be determined before consume the capsule with pterostilbene until 24 hours postprandially at 8 points after consuming the capsule (0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours and 24 hours).
Relative oral bioavailability (Frel) | At week 1 and week 2
  Fasting pterostilbene levels in plasma will be determined before consume the capsule with pterostilbene until 24 hours postprandially at 8 points after consuming the capsule (0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours and 24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — UTNS (Eurecat_Reus)
Locations (1):
- Eurecat, Reus, Spain

IPD SHARING:
Plan to Share IPD: No
In this study IPD will not be shared with other researchers because all the information will be processed by the UTNS of Eurecat.

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org